CLINICAL TRIAL: NCT01812226
Title: Alcohol Biomarkers in Post-Liver Transplant Patients
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Michael Fleming, Professor, Northwestern University
Other Study IDs: STU31235
Record Dates: First submitted 2013-03-11; First posted 2013-03-18 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Alcohol-related Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected to detect PEth levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- experimental group: This group will consist of men and women who received a liver transplant for alcohol-related liver disease.
- control group: This group will consist of men and women who had a liver transplant for reasons that are not alcohol-related.

SUMMARY:
The aim of this study is to compare the predictive validity and reliability of PEth testing at detecting alcohol use in post liver transplant patients. A prospective cohort study will be used to test the primary hypothesis. Subjects enrolled in the study will be followed for 12 months with biomarker levels drawn at baseline, six and 12 months. The baseline interview will inquire about the previous 30 day alcohol and tobacco use; lifetime and 12 month Diagnostic and Statistical Manual-IV criteria for alcohol abuse and/or dependence; prior alcohol treatment; history of abstinence prior to transplant; co-morbid medical issues; and depression. The six and 12 months interview will focus on previous 30 day alcohol use. The baseline, six and 12 months interviews will be conducted face-to-face at each site. While many patients who receive a transplant do not live near the academic medical center that performed the surgery patient, they normally have a transplant clinic visit 1-2 times per year. Medical records and transplant databases will be assessed to assess the other variables of interest.

DETAILED DESCRIPTION:
Patients who have a positive PEth will be asked to have a confirmatory test performed 10-14 days after a positive result (PEth >20ng/ml). The rationale for this procedure is to determine the test retest reliability of this marker and as well as being able to correlate levels of drinking with changes in biomarker levels over time. There is limited information on the length of time PEth levels remain elevated in transplant patients after drinking episodes.

Hypothesis H.1. PEth will have a significantly higher "area under the Receiver Operating Characteristic (ROC) curve" in a sample of post-transplant patients who report any alcohol use in the past 30 days compared to the control group.

H.2. PEth will have a significantly higher "area under the ROC curve" in a sample of post-transplant patients who report daily alcohol use of >40 grams/day (three drinks/day) in the past 30 days compared to the control group.

H.3. PEth will have a significantly higher "area under the ROC curve" in a sample of post-transplant patients who report heavy episodic drinking (>60 grams of alcohol, eight or more occasions in the past 30 days) compared to the control group.

H.4. PEth levels will be <20 ng/ml in the control sample of 50 post transplant patients who do not have a history of alcohol dependence or alcohol related liver disease.

H.5. The test-retest reliability of PEth will be >0.90.

ELIGIBILITY:
Inclusion Criteria:

* men and women 18 years and over
* Participant must have received a liver transplant after January 1, 2003
* Participant must be six months or more post-transplant
* Mini-mental status score of greater than or equal to 20
* Participant must be well enough to participate in the research procedures over a 12 month period
* Participant must continue to be followed by the transplant center

Exclusion Criteria:

* Individuals who do not consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transplant center patients
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2013-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
specificity of PEth to detect alcohol use among post-transplant patients | 12 month follow up
  The criteria standard on which we will base the specificity will be a combination of patient self-report, family member report and clinician/medical record data.
  Subjects in whom any concern of current alcohol use, from any of these sources, would be considered a positive for current drinking.
  The PEth levels would then be compared to this standard of current alcohol use
  Data from previous research suggests PEth has a specificity close to 100%

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Fleming, MD, MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Wisconsin, Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No